CLINICAL TRIAL: NCT04035018
Title: A Study on the Effectiveness of Pharmacopuncture for Chronic Neck Pain: A Protocol for a Pragmatic Randomized Controlled Trial
Brief Title: Effectiveness of Pharmacopuncture for Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2019-04
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Chronic Neck Pain
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pharmacopuncture therapy (Experimental): The physicians will select one or more pharmacopuncture therapy for each participants. The physicians will also decide dosage and frequency of treatment according to the participant's status.
  Interventions: Procedure: pharmacopuncture therapy
- physical therapy (Active Comparator): The physicians will select one or more physical therapy for each participants. The physicians will also decide intensity and frequency of treatment according to the participant's status.
  Interventions: Procedure: Physical therapy

INTERVENTIONS:
Procedure: pharmacopuncture therapy — The participants in the treatment group will be receive one or more pharmacopuncture therapy according to the physician's decision.
  Arms: pharmacopuncture therapy
Procedure: Physical therapy — The participants in the control group will be receive one or more physical therapy according to the physician's decision.
  Arms: physical therapy

SUMMARY:
In this study, the investigators will evaluate the efficacy and safety of pharmacopuncture therapy for chronic neck pain compared to physical therapy.

DETAILED DESCRIPTION:
This study is prgmatic RCT of pharmacopuncture therapy for chronic neck pain compared to physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain more than 6 months
* VAS of neck pain more than 5
* Age between 17 and 70 years old
* Participants who wrote informed consent

Exclusion Criteria:

* Migration of cancer reaching to spine, fracture of spine
* Progressive neurologic deficits or severe neurologic deficits
* Cancer, fibromyalgia, RA, or goat
* Stroke, MI, kidney disease, dimentia, diabetic neuropathy, or epilepsy
* Participants taking steroid, immunosuppressant, or psychotropic medication
* Hemorrhagic disease, severe diabetes or taking anticoagulant drug
* Participants who took NSAIDs or pharmacopuncture within 1 week
* Pregnant or lactating women
* Participants who had undergone cervical surgery within 3 months
* Participants who had participated in other clinical trial within 1 month, or have plan for participation in other trial during follow up period of this trial
* Participants who can not write informed consent
* Participants who is difficult to participate in the trial according to investigator's decision

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale of neck pain | week 6
  Minimum 0, Maximum 100. Higher values represent a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Principal Investigator — Jaseng Hospital of Korean Medicine
Locations (4):
- South Korea (4):
  - Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi Province
  - Haeundae Jaseng Hospital of Korean Medicine, Busan
  - Daejeon Jaseng Hospital of Korean Medicine, Daejeon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SM, Kim SJ, Nam D, Park YC, Kim EJ, Ha IH, Lee YJ. Comparison of preference-based health-related quality of life measures for chronic neck pain: a pooled analysis of data from three RCTs. BMJ Open. 2024 Dec 26;14(12):e086104. doi: 10.1136/bmjopen-2024-086104. PMID 39725423
- [Derived] Kim D, Kim ES, Song HJ, Park SY, Park KS, Lee YJ, Ha IH. An economic evaluation of pharmacopuncture versus usual care for chronic neck pain: a pragmatic randomized controlled trial. BMC Health Serv Res. 2023 Nov 23;23(1):1286. doi: 10.1186/s12913-023-10325-w. PMID 37993844
- [Derived] Park KS, Kim S, Kim C, Seo JY, Cho H, Kim SD, Lee YJ, Lee J, Ha IH. A Comparative Study of the Effectiveness of Pharmacopuncture Therapy for Chronic Neck Pain: A Pragmatic, Randomized, Controlled Trial. J Clin Med. 2021 Dec 21;11(1):12. doi: 10.3390/jcm11010012. PMID 35011752